CLINICAL TRIAL: NCT04376697
Title: Repetitive Transcranial Magnetic Stimulation Trajectory of Outcomes Study in Major Depression
Brief Title: Repetitive Transcranial Magnetic Stimulation Trajectory of Outcomes Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Jonathan Downar, Clinician scientist, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-6253.1
Record Dates: First submitted 2020-04-25; First posted 2020-05-06 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Depressive Disorder
Keywords: rTMS; TMS; repetitive transcranial magnetic stimulation; major depressive disorder; major depression; MDD
MeSH Terms: conditions — Depressive Disorder; Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: prospective, single-arm, open label feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active rTMS (Experimental): Treatment will be delivered daily (weekdays) rTMS treatments, for up to 10 daily sessions and up to 75 sessions in total.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — The treatment will be delivered by trained medical personnel.

SUMMARY:
This prospective, single-arm, open-label feasibility study will assess the safety, tolerability, and effectiveness of repetitive transcranial magnetic stimulation (rTMS) in patients with major depression (MDD) to test the hypothesis that remission rates can be increased by additional treatment sessions.

ELIGIBILITY:
Inclusion Criteria:

* are outpatients
* are voluntary and competent to consent to treatment
* are between the ages of 18 and 85, inclusive
* are able to adhere to the treatment schedule
* pass the TMS safety-screening questionnaire
* have had no change or initiation of any psychotropic medication in the 4 weeks prior to screening

Exclusion Criteria:

* previous rTMS treatment
* have a history of substance dependence or abuse within the last 3 months
* have a concomitant major unstable medical illness, cardiac pacemaker or implanted medication pump
* have active suicidal intent
* have a diagnosis of any personality disorder, and assessed by a study investigator to be primary and causing greater impairment than MDD
* have a diagnosis of any psychotic disorder
* have any significant neurological disorder or insult including, but not limited to: any condition likely to be associated with increased intracranial pressure, space occupying brain lesion, any history of seizure confirmed diagnostically by neurological assessment (except those therapeutically induced by ECT), cerebral aneurysm, Parkinson's disease, Huntington's chorea, dementia, stroke, neurologically confirmed diagnosis of traumatic brain injury, or multiple sclerosis.
* if participating in psychotherapy, must have been in stable treatment for at least 3 months prior to entry into the study, with no anticipation of change in the frequency of therapeutic sessions, or the therapeutic focus over the duration of the study
* clinically significant laboratory abnormality, in the opinion of the investigator
* currently (or in the last 4 weeks) take more than lorazepam 4 mg daily (or equivalent) or any dose of an anticonvulsant due to the potential to limit rTMS efficacy
* non-correctable clinically significant sensory impairment (i.e., cannot hear well enough to cooperate with interview)
* any significant cardiovascular or metabolic disorder or insult including, but not limited to: coronary artery disease, abnormal heart rhythms, heart failure, cardiac valve disease, congenital heart disease, cardiomyopathy, vascular disease, dyslipidemia, diabetes, or hypertension

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-03-18 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Beck Depression Inventory-II (BDI-II) (score 0-63, higher = more severe) | Baseline (week prior to treatment), on each treatment day, 1 week and 4 weeks post-treatment
  Outcome measured by a change in depression score at baseline, before every treatment, and at 1 and 4 weeks post-treatment. A 50% improvement in the score is considered a response to rTMS. A score of 12 or less is categorized as remission.

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale 17-items (HDRS17) (score 0-52, higher = more severe) | Baseline (week prior to treatment) and after 1 week and 4 weeks post-treatment
  Outcome measured by a change in depression score from baseline (week prior to treatment) to 1 week and 4 weeks post-treatment. A 50% improvement in the score is considered a response to rTMS. A score of 7 or less is categorized as remission.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Downar, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sheen JZ, Miron JP, Mansouri F, Dunlop K, Russell T, Zhou R, Hyde M, Fox L, Voetterl H, Daskalakis ZJ, Griffiths JD, Blumberger DM, Downar J. Cardiovascular biomarkers of response to accelerated low frequency repetitive transcranial magnetic stimulation in major depression. J Affect Disord. 2022 Dec 1;318:167-174. doi: 10.1016/j.jad.2022.08.105. Epub 2022 Aug 31. PMID 36055538
- [Derived] Miron JP, Voetterl H, Fox L, Hyde M, Mansouri F, Dees S, Zhou R, Sheen J, Desbeaumes Jodoin V, Mir-Moghtadaei A, Blumberger DM, Daskalakis ZJ, Vila-Rodriguez F, Downar J. Optimized repetitive transcranial magnetic stimulation techniques for the treatment of major depression: A proof of concept study. Psychiatry Res. 2021 Apr;298:113790. doi: 10.1016/j.psychres.2021.113790. Epub 2021 Feb 7. PMID 33581379